CLINICAL TRIAL: NCT01327183
Title: A MULTI-CENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY EVALUATING THE EFFICACY AND SAFETY OF 2 DOSES OF RO4905417 (R1512) ADMINISTERED TO PATIENTS WITH NON ST-ELEVATION MYOCARDIAL INFARCTION (NON-STEMI) UNDERGOING PERCUTANEOUS CORONARY INTERVENTION (PCI)
Brief Title: A Study of RO4905417 in Patients With Non ST-Elevation Myocardial Infarction (Non-STEMI) Undergoing Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP25619
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Percutaneous Coronary Intervention; inclacumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 20 mg/kg RO4905417 before PCI (Experimental)
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI); Drug: RO4905417
- 5 mg/kg RO4905417 before PCI (Experimental)
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI); Drug: RO4905417
- Placebo before PCI (Placebo Comparator)
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI); Drug: placebo

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention (PCI) — at least 1 hour and up to 24 hours after completion of drug infusion
Drug: RO4905417 — 5 mg/kg iv infusion, completed at least 1 hour and up to 24 hours before PCI
  Arms: 5 mg/kg RO4905417 before PCI
Drug: RO4905417 — 20 mg/kg iv infusion, completed at least 1 hour and up to 24 hours before PCI
  Arms: 20 mg/kg RO4905417 before PCI
Drug: placebo — iv infusion, completed at least 1 hour and up to 24 hours before PCI
  Arms: Placebo before PCI

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of RO4905417 in patients with non ST-elevation myocardial infarction (Non-STEMI) undergoing percutaneous coronary intervention (PCI). Patients will be randomized to receive an intravenous infusion of either 5 mg/kg RO4905417 or 20 mg/kg RO4905417 or placebo before PCI. Follow-up will be for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >18 to <75 years of age
* Non ST-elevation myocardial infarction
* Woman of childbearing potential will be allowed only if using two acceptable methods of contraception
* Body mass index (BMI) </= 40 kg/m2

Exclusion Criteria:

* Acute ST-elevation myocardial infarction (STEMI)
* Culprit coronary lesion with a total thrombotic occlusion or a lesion requiring the use of distal embolization protection or thrombectomy devices
* Percutaneous coronary intervention (PCI) within the past 72 hours
* Thrombolytic therapy within the past 7 days
* Major surgery within the past 3 months
* History of cerebral vascular disease or stroke in the past 3 months
* Bleeding disorders
* Inadequately controlled severe hypertension
* Prior coronary artery bypass graft (CABG) surgery
* Decompensated heart failure (oedema and/or rale)
* Acute infection at screening or active chronic infection within 3 months prior to PCI
* Patients known to be HIV positive, patients receiving antiretroviral drugs, or immuno-suppressed patients
* Uncontrolled diabetes mellitus (HbA1C >10%) at baseline

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Reduction of procedural damage during percutaneous coronary intervention (PCI): Change from baseline in troponin I levels early after PCI | from baseline to 24 hours post PCI

SECONDARY OUTCOMES:
Change from baseline in troponin I at 8 hours post PCI | from baseline to 8 hours post PCI
Peak and AUC for troponin I | 24 hours post PCI
Change from baseline in Creatine Kinase-Myocardial Band (CK-MB) after PCI | from baseline to 24 hours post PCI
Change form baseline in Growth Differentiation Factor 15 (GDF-15) at 120 days post PCI | from baseline to Day 120 post PCI
Change from baseline in cystatin C biomarker at 24 hours and 30 days post PCI | from baseline to Day 30 post PCI
Safety: Incidence of adverse events and major adverse cardiovascular events (MACEs) | 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (61):
- United States (34):
  - Huntsville, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - Salinas, California
  - Littleton, Colorado
  - Farmington, Connecticut
  - Boynton Beach, Florida
  - Kissimmee, Florida
  - Ocala, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Columbus, Georgia
  - Aurora, Illinois
  - Fort Wayne, Indiana
  - Iowa City, Iowa
  - Wichita, Kansas
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Baltimore, Massachusetts
  - Hyannis, Massachusetts
  - Bay City, Michigan
  - Petoskey, Michigan
  - Saint Paul, Minnesota
  - Ridgewood, New Jersey
  - Johnson City, New York
  - Raleigh, North Carolina
  - Bismarck, North Dakota
  - Springfield, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Chambersburg, Pennsylvania
  - Houston, Texas
- Canada (10):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Hamilton, Ontario
  - Newmarket, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Charles-Borromée, Quebec
- Netherlands (5):
  - Heerlen
  - Leeuwarden
  - Nijmegen
  - Rotterdam
  - Tilburg
- Poland (12):
  - Bydgoszcz
  - Gdansk
  - Gdynia
  - Józefów
  - Katowice
  - Krakow
  - Lodz
  - Starogard Gdański
  - Torun
  - Warsaw
  - Wejherowo
  - Wroclaw

REFERENCES:
- [Derived] Stahli BE, Gebhard C, Duchatelle V, Cournoyer D, Petroni T, Tanguay JF, Robb S, Mann J, Guertin MC, Wright RS, L L'Allier P, Tardif JC. Effects of the P-Selectin Antagonist Inclacumab on Myocardial Damage After Percutaneous Coronary Intervention According to Timing of Infusion: Insights From the SELECT-ACS Trial. J Am Heart Assoc. 2016 Nov 16;5(11):e004255. doi: 10.1161/JAHA.116.004255. PMID 27852589
- [Derived] Tardif JC, Tanguay JF, Wright SR, Duchatelle V, Petroni T, Gregoire JC, Ibrahim R, Heinonen TM, Robb S, Bertrand OF, Cournoyer D, Johnson D, Mann J, Guertin MC, L'Allier PL. Effects of the P-selectin antagonist inclacumab on myocardial damage after percutaneous coronary intervention for non-ST-segment elevation myocardial infarction: results of the SELECT-ACS trial. J Am Coll Cardiol. 2013 May 21;61(20):2048-55. doi: 10.1016/j.jacc.2013.03.003. Epub 2013 Mar 10. PMID 23500230